CLINICAL TRIAL: NCT06038032
Title: The RESILIENCE Trial: Using a Multimodal and Digital Intervention to Optimize Waist Circumference, Body Composition, and Cardiometabolic Health in Endometrial Cancer Survivors.
Brief Title: ImpRoving hEalth behaviourS for LIfe After ENdometrial CancEr Trial
Acronym: RESILIENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-23-0209
Record Dates: First submitted 2023-08-24; First posted 2023-09-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive the intervention for 24 weeks. The first 16 weeks will involve an intensive behavioral program (digital wellness platform plus online healthcare professional support), followed by an 8-week maintenance period (digital wellness platform alone).
  At baseline, participants will receive handouts with publicly available health information; they will also wear an activity monitor and receive support telephone calls for the 24 weeks.
  Interventions: Behavioral: Digital wellness platform; Behavioral: Online healthcare professional support
- Control group (No Intervention): At baseline, participants will receive handouts with publicly available health information; they will also wear an activity monitor and receive support telephone calls for the 24 weeks.

INTERVENTIONS:
Behavioral: Digital wellness platform — A digital wellness platform based on preventive self-care that contains tools to monitor nutrition, physical activity, and mental wellbeing will be accessed daily for 24 weeks.
  Arms: Intervention group
Behavioral: Online healthcare professional support — Individual sessions with a registered dietitian, an exercise professional, and a mental health therapist for 16 weeks.
  Arms: Intervention group

SUMMARY:
RESILIENCE is 24-week randomized controlled trial that assesses the efficacy of a digital wellness platform, combined with online support from healthcare professionals, to enhance waist circumference and other vital health outcomes in endometrial cancer survivors.

DETAILED DESCRIPTION:
Background: Individuals diagnosed with endometrial cancer are at an increased risk of cardiac complications post-treatment, particularly if having overweight or a pronounced waist size. Adopting healthy habits-like nutritious eating, regular physical activity, and effective stress management-can mitigate these risks and bolster overall health. However, many cancer survivors find it challenging to consistently adhere to these health and wellness recommendations.

Objective: This study aims to determine the efficacy of a digital wellness platform, enriched with professional guidance, in facilitating healthier lifestyles for endometrial cancer survivors. This would encompass enhancements in nutrition, physical activity levels, and mindfulness practices.

Study Design:

Group 1 (Intervention Group): Participants will engage with the digital wellness platform daily for the initial 16 weeks with expert guidance. Subsequently, participants will navigate the platform independently for the next 8 weeks.

Group 2 (Control Group): Participants will initially be provided with standard publicly accessible health information. After the primary 24-week period, participants will gain access to the digital wellness platform.

Common Elements: Both groups will have access to general health information and will benefit from supportive calls. To monitor their physical activity, all participants will be equipped with an activity tracker.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Histologically confirmed endometrioid adenocarcinoma (low-grade), FIGO 2009 stages I to III.
* 1 month to 10 years post-surgery and completion of adjuvant treatment.
* BMI ≥25 and ≤45 kg/m2.
* Willing and able to adhere to the study interventions and assessments
* Seeking best weight using the readiness to change questionnaire.
* Have a cell phone compatible with the Fitbit app with internet access and Bluetooth capabilities.
* Able to speak, read and understand English.

Exclusion Criteria:

* Recurrent (local, regional, or distant) or metastatic EC.
* Abnormal (i.e., mutated) p53 status in combination with FIGO 2009 stage III or IV
* Weight fluctuations (±5 kg) within the previous 3 months.
* Planned surgery in the next 6 months.
* Previous bariatric surgery.
* Uncontrolled thyroid disorder
* Type 1 diabetes.
* Type 2 diabetes with HbA1c > 10% or are taking insulin, sulfonylureas, or GLP-1 agonists.
* Taking corticosteroids.
* Taking anti-obesity drugs.
* Current smoker (of any type, e.g e-cigarettes, tobacco, marihuana, vaping)
* Self-report >90 moderate-intensity min/week of aerobic physical activity on average over the past three months.
* Potential safety risk with exercise or maximal exercise testing screened with the 2023 Physical Activity Readiness Questionnaire (PAR-Q+)53, signs and symptoms of CVD, and any of the American Heart Association's absolute or relative contraindications to exercise testing.
* Physical or mobility limitations impacting ability to perform physical activity.
* Self-report following a structured hypocaloric diet (e.g., using formulated meal replacements, weight loss meal program) or a restrictive diet (intermittent fasting, or high-fat diet) in the past three months, or self-report currently following a vegan diet but for less than two years.
* Self-reported history of an eating disorder diagnosed by a physician.
* Intending to be away longer than 2 weeks consecutively during the intervention and unable to adhere to the study protocol during this period.
* Active substance abuse (alcohol, cannabis, illicit drugs, prescription drugs).
* Dual-energy x-ray absorptiometry (DXA) or magnetic resonance imaging (MRI) contraindications for research purposes, such as pacemakers or pregnancy
* Unable to participate in telephone and virtual intervention protocols (e.g., having a severe hearing or vision loss).
* Unable to adhere to the study protocol (i.e., unavailable to commit to scheduled group video conferencing sessions; limited access to the Internet; not willing to use platform, individuals who have been advised by a health professional not to lose weight or reduce caloric intake; cognitive impairment or dementia; etc.).
* Unable to come to study location.
* Unable to provide written informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in waist circumference at week 16. | Baseline to week 16
  Waist circumference will be measured in centimeters (cm) using an inelastic tape at the level of the iliac crest at the end of normal expiration.

SECONDARY OUTCOMES:
Change from baseline in waist circumference at week 24. | Baseline and week 24
  Waist circumference will be measured in centimeters (cm) using an inelastic tape at the level of the iliac crest at the end of normal expiration.
Change from baseline in body weight (in kg) at weeks 16 and 24. | Baseline, week 16, and week 24
  Weight will be measured in kilograms (kg) in triplicate following standardized procedures; average values will be used for analysis.
Change from baseline in fat mass by DXA at weeks 16 and 24. | Baseline, week 16, and week 24
  Percentage fat mass will be measured using dual-energy x-ray absorptiometry (DXA), which is a precise and reliable technique.
Change from baseline in appendicular lean soft tissue by DXA at weeks 16 and 24. | Baseline, week 16, and week 24
  Appendicular lean soft tissue will be measured using dual-energy x-ray absorptiometry (DXA), which is a precise and reliable technique. Appendicular lean soft tissue will be adjusted for body weight.
Change from baseline in metabolic syndrome by Z score calculation at weeks 16 and 24. | Baseline, week 16, and week 24
  Metabolic syndrome severity Z score will be calculated using waist circumference, blood pressure, high-density lipoprotein cholesterol, triglycerides, and fasting glucose data in sex- and ethnicity-specific equations.
Change from baseline in cardiovascular risk based on the Framingham risk score at weeks 16 and 24. | Baseline, week 16, and week 24
  10-year cardiovascular risk will be estimated using sex-specific Framingham risk score based on traditional risk factors. Risk is low if the score is less than 10% and high if it is 20% or higher.
Change from baseline in handgrip muscle strength at weeks 16 and 24. | Baseline, week 16, and week 24
  Handgrip strength will be evaluated using a hydraulic handgrip dynamometer.
Change from baseline in cardiorespiratory fitness by a cardiopulmonary exercise testing (CPET) at weeks 16 and 24. | Baseline, week 16, and week 24
  Peak oxygen uptake will be measured by gold standard cardiopulmonary exercise testing.
Change from baseline in health-related life improvement by the QLQ-C30 at weeks 16 and 24. | Baseline, week 16, and week 24
  Participants will complete the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core-30 (QLQ-C30). Score ranges from 0 to 100. Higher scores on symptoms and single-items indicate a higher level of symptoms.
Change from baseline in health-related life improvement by the QLQ-EN24 at weeks 16 and 24. | Baseline, week 16, and week 24
  Participants will complete the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire -Endometrial Cancer Module (EORTC QLQ-EN24). Score ranges from 0 to 100. Higher scores on symptoms and single-items indicate a higher level of symptoms.
Change from baseline in carotid intima-media thickness by ultrasound at weeks 16 and 24. | Baseline, week 16, and week 24
  Carotid intima-media thickness will be assessed by a B-mode ultrasound following a standardized protocol.
Change from baseline in abdominal adiposity by MRI at week 24. | Baseline and week 24
  Abdominal adipose tissue will be measure using magnetic resonance imaging (MRI).
Change from baseline in abdominal skeletal muscle by MRI at week 24. | Baseline and week 24
  Abdominal skeletal muscle will be measure using magnetic resonance imaging (MRI).
Change from baseline in adipose tissue in liver by MRI at week 24. | Baseline and week 24
  Adipose tissue in liver will be measure using magnetic resonance imaging (MRI).
Change from baseline in adipose tissue in the thigh region by MRI at week 24. | Baseline and week 24
  Adipose tissue in the thigh region will be measure using magnetic resonance imaging (MRI).
Change from baseline in skeletal muscle in the thigh region by MRI at week 24. | Baseline and week 24
  Skeletal muscle in the thigh region will be measure using magnetic resonance imaging (MRI).
Change from baseline in cardiac function by MRI at week 24. | Baseline and week 24
  Cardiac function will be measure using magnetic resonance imaging (MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Carla Prado, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of Toronto, Toronto

IPD SHARING:
Plan to Share IPD: No